CLINICAL TRIAL: NCT04144517
Title: A Phase 2 Study of ALKS 4230 in Combination With Anti-PD-1 (Pembrolizumab) in Patients With Advanced or Recurrent Head and Neck Squamous Cell Cancer Currently on Treatment With Anti-PD-(L)1 Without Having Achieved a Complete Remission
Brief Title: A Study of ALKS 4230 (Nemvaleukin Alfa) With Pembrolizumab in Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mural Oncology, Inc (Industry)
Collaborators: Immune Oncology Network (ION) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ION-01-ALKS 4230
Record Dates: First submitted 2019-10-24; First posted 2019-10-30 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Alkermes; IL-2; Interleukin-2; Oncology; Immuno-oncology; Cytokine Immunotherapy; ALKS 4230; Pembrolizumab; Keytruda; PD-L1; Solid Tumors
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Nemvaleukin 3 mcg/kg + Pembrolizumab 200 mg (Experimental): Participants with current stable disease (SD) or partial response (PR) (Cohorts 1 and 2) who were not progressing or further demonstrating reductions in tumor size were to receive nemvaleukin alfa 3 microgram per kilogram (mcg/kg), intravenous (IV) infusion, daily from Days 1 to 5 of the first week of each 3-week treatment cycle in combination with pembrolizumab 200 milligram (mg), IV infusion, once, every three weeks (Q3W) on Day 1 of each 21-day cycle until confirmed progression, unacceptable toxicity or met other criteria for discontinuation.
  Interventions: Drug: Nemvaleukin Alfa; Drug: Pembrolizumab
- Group 2: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg (Experimental): Participants with progressive disease (PD) (Cohorts 3 and 4) received nemvaleukin alfa 3 mcg/kg, IV infusion, daily from Days 1 to 5 of the first week of each 3-week treatment cycle in combination with pembrolizumab 200 mg, IV infusion, once, Q3W on Day 1 of each 21-day cycle until confirmed progression, unacceptable toxicity or met other criteria for discontinuation.
  Interventions: Drug: Nemvaleukin Alfa; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Nemvaleukin Alfa — Nemvaleukin alfa IV infusion.
Drug: Pembrolizumab — Pembrolizumab IV infusion.
  Other Names: Keytruda

SUMMARY:
The primary objective of this study was to estimate the response rate to ALKS 4230 in combination with pembrolizumab in patients with HNSCC who had previously received anti-PD-(L)1 therapy but who had not achieved a CR.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytopathologically confirmed diagnosis of non-cutaneous squamous cell carcinoma of the head and neck region that is locally advanced and/or recurrent and no longer amenable to local surgical or radiation therapy and/or with evidence of distant metastatic disease
* Patients must have had anti-PD-(L)1 therapy as the most recent systemic therapy with either stable disease or partial response on prior anti-PD-(L)1 therapy, or progressive disease on prior anti-PD-(L)1 therapy
* Patients must have disease that is measurable by RECIST v1.1
* Patients must be willing to provide tumor tissue biopsy
* Patients must demonstrate adequate organ function
* Female patients of childbearing potential should have a negative pregnancy test within 72 hours prior to receiving the first dose of study medication
* Patients must agree to follow contraceptive requirements defined in the protocol
* Additional criteria apply

Exclusion Criteria:

* Patient is pregnant or breastfeeding or expecting to conceive or father children
* Patient has an active major infection requiring systemic therapy within 1 week of starting study drug
* Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate, provided that they are stable, have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study drug
* Patient has hypersensitivity to pembrolizumab, ALKS 4230, or any of their excipients
* Patient has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (inhaled or topical steroids and steroid replacement at physiologic doses are allowable)
* Patient has prior Grade ≥3 immune-related toxicities requiring systemic immunosuppressant treatment that were attributable or possibly attributable to PD-1 immune checkpoint blockade
* Patient has active tuberculosis or known active infection with hepatitis B or hepatitis C
* Patient has known psychiatric or substance abuse disorders or a social situation that would interfere with cooperation with the requirements of the study
* Additional criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2022-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Mural Oncology, Inc
Locations (6):
- United States (6):
  - Mural Oncology Investigational Site, Miami, Florida
  - Mural Oncology Investigational Site, Atlanta, Georgia
  - Mural Oncology Investigational Site, Minneapolis, Minnesota
  - Mural Oncology Investigational Site, New York, New York
  - Mural Oncology Investigational Site, Cleveland, Ohio
  - Mural Oncology Investigational Site, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in the United States.
Pre-assignment Details: This study consisted of Group 1 (Cohorts 1 and 2) and Group 2 (Cohorts 3 and 4). Group 1 was closed due to lack of recruitment of eligible participants and therefore, no data for Group 1 (Cohorts 1 and 2) were collected, analyzed or reported. Data was collected and analyzed for Group 2 and is presented in this results report.
Groups:
- Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg: Participants with advanced, recurrent and/or metastatic squamous cell carcinoma of the head and neck (HNSCC) and with progressive disease (PD) with no prior response to greater than or equal to (>=) 8 weeks anti programmed cell death ligand-1 (anti-PD-[L]1) therapy received nemvaleukin alfa 3 microgram per kilogram (mcg/kg), intravenous (IV) infusion, daily from Days 1 to 5 of the first week of each 3-week treatment cycle in combination with pembrolizumab 200 milligram (mg), IV infusion, once, every three weeks (Q3W) on Day 1 of each 21-day cycle until confirmed progression, unacceptable toxicity or met other criteria for discontinuation.
- Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg: Participants with advanced, recurrent and/or metastatic HNSCC and with current PD after prior achievement of best response stable disease (SD) or partial response (PR) and after >=8 on weeks on anti-PD-(L)1 therapy received nemvaleukin alfa 3 mcg/kg, IV infusion, daily from Days 1 to 5 of the first week of each 3-week treatment cycle in combination with pembrolizumab 200 mg, IV infusion, once, Q3W on Day 1 of each 21-day cycle until confirmed progression, unacceptable toxicity or met other criteria for discontinuation.
Period: Overall Study
Arm/Group | Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg
Started | 8 | 6
Completed | 0 | 0
Not Completed | 8 | 6
Not completed — Physician Decision | 0 | 1
Not completed — Other | 2 | 2
Not completed — Death | 6 | 3

BASELINE CHARACTERISTICS:
Population: Safety population included participants who received at least one dose of either study drug (nemvaleukin alfa or pembrolizumab).
Groups:
- Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg: Participants with advanced, recurrent and/or metastatic squamous cell carcinoma of the HNSCC and with PD with no prior response to >=8 weeks anti-PD-(L)1) therapy received nemvaleukin alfa 3 mcg/kg, IV infusion, daily from Days 1 to 5 of the first week of each 3-week treatment cycle in combination with pembrolizumab 200 mg, IV infusion, once, Q3W on Day 1 of each 21-day cycle until confirmed progression, unacceptable toxicity or met other criteria for discontinuation.
- Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg: Participants with advanced, recurrent and/or metastatic HNSCC and with current PD after prior achievement of best response SD or PR and after >=8 on weeks on anti-PD-(L)1 therapy received nemvaleukin alfa 3 mcg/kg, IV infusion, daily from Days 1 to 5 of the first week of each 3-week treatment cycle in combination with pembrolizumab 200 mg, IV infusion, once, Q3W on Day 1 of each 21-day cycle until confirmed progression, unacceptable toxicity or met other criteria for discontinuation.
- Total: Total of all reporting groups
Arm/Group | Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (15.19) | 62.3 (8.62) | 62.3 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Based on RECIST v1.1
Description: ORR was defined as percentage of participants with complete response (CR) or PR as assessed by investigator based on response evaluation criteria in solid tumors (RECIST) version (v) 1.1. CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis less than (<) 10 millimeters (mm). PR was defined as at least a 30 percent (%) decrease in the sum of diameter (SOD) of target lesions, taking as reference the baseline sum diameters. PD was defined as at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From the first dose of study drug until first PD or death, whichever occurred first (up to 49 weeks)
Population: Efficacy evaluable population included all participants who received at least one dose of both study drugs (nemvaleukin alfa or pembrolizumab) and had measurable disease at post-baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 8 | 6
percentage of participants | 0 [NA to NA] — Upper and lower limit of 95% Confidence interval (CI) could not be estimated due to insufficient participants with events. | 16.7 [0.4 to 64.1]

2. Secondary Outcome: Duration of Response (DOR) Based on RECIST v1.1
Description: DOR was defined as time in months from the first documentation CR or PR until the first documentation of confirmed PD as assessed by investigator based on RECIST v1.1. CR: disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis <10 mm. PR: at least a 30% decrease in the SOD of target lesions, taking as reference the baseline sum diameters. PD: at least 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the smallest sum and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: From first documented CR or PR until first documentation of PD (up to 49 weeks)
Population: Efficacy evaluable population included all participants who received at least one dose of both study drugs (nemvaleukin alfa or pembrolizumab) and had measurable disease at post-baseline. Here, 'overall number of participants analyzed' signifies participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 0 | 1
months |  | NA [NA to NA] — Median and upper and lower limit of 95% CI could not be estimated due to insufficient participants with events.

3. Secondary Outcome: Progression-free Survival (PFS) Based on RECIST v1.1
Description: PFS was defined as the time (in months) from the date of first dose of study drug to the date of first documentation of objective tumor progression, start of alternate therapy or death due to any cause, whichever occurred first, based on RECIST v1.1. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the baseline SOD of target lesions.
Time Frame: From the first dose of study drug to date of PD, start of alternate therapy or death, whichever occurred first (up to 49 weeks)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 8 | 6
months | 1.3 [1.1 to 1.5] | NA [1.2 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient events.

4. Secondary Outcome: Time to Progression (TTP) Based on RECIST v1.1
Description: TTP was defined as the time from the date of first dose of study drug to the date of first documentation of PD based on RECIST 1.1. PD was defined as at least a 20% increase (including an absolute increase of at least 5 mm) in the SOD of target lesions, taking as reference the baseline SOD of target lesions.
Time Frame: From first dose of study drug to the date of the first documentation of PD (up to 49 weeks)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 8 | 6
months | 1.3 [1.1 to 1.5] | NA [1.2 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient events.

5. Secondary Outcome: Disease Control Rate (DCR) Based on RECIST v1.1
Description: DCR was defined as percentage participants with a confirmed CR, PR, or SD as assessed by an investigator based on RECIST v1.1. CR: disappearance of all target lesions. All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to <10 mm. PR: at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameter. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study (this includes baseline sum if that is the smallest on study).
Time Frame: From first dose of study drug until PD or death, whichever occurred first (up to 49 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 8 | 6
percentage of participants | 12.5 [0.3 to 52.7] | 83.3 [35.9 to 99.6]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose of study drug until the date of death due to any cause. Participants were followed for survival after the last dose of study drug.
Time Frame: From date of first dose of study drug up to death from any cause (up to 89 weeks)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 8 | 6
months | 5.4 [1.8 to NA] — Upper limit of 95% CI could not be estimated due to insufficient events. | NA [3.9 to NA] — Median and upper limit of 95% CI could not be estimated due to insufficient events.

7. Secondary Outcome: Number of Participants With Drug-related Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant who was administered a pharmaceutical product. A SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required participant's hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, led to a congenital anomaly/birth defect. TEAE included AE that occurred or worsen after the first dose of study drug. The assessment of the relationship of study drug to TEAEs and SAEs was done by the Investigator (or designated sub-Investigator) according to their best clinical judgment.
Time Frame: From the first dose of study drug through 90 days after the last dose of study drug (up to 62 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 8 | 6
Participants
  Nemvaleukin Alfa Related TEAEs | 6 | 4
  Pembrolizumab Related TEAEs | 4 | 4
  Nemvaleukin Alfa Related SAEs | 0 | 1
  Pembrolizumab Related SAEs | 0 | 1

8. Secondary Outcome: Number of Participants With Drug-related TEAEs Leading to Discontinuation of Treatment
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant who was administered a pharmaceutical product. TEAE included AE that occurred or worsen after the first dose of study drug. The assessment of the relationship of study drug to AEs was done by the Investigator (or designated sub-Investigator) according to their best clinical judgment.
Time Frame: From first dose of study drug through 90 days after the last dose of study drug (up to 62 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg
Number analyzed (Participants) | 8 | 6
Participants
  Participants With Drug-related TEAEs Leading to Discontinuation of Nemvaleukin Alfa | 3 | 0
  Participants With Drug-related TEAEs Leading to Discontinuation of Pembrolizumab | 3 | 0

ADVERSE EVENTS:
Time Frame: Serious and Other (non-serious) AEs: From the first dose of study drug through 90 days after the last dose of study drug (up to 62 weeks); Mortality: From first dose of study drug up to 89 weeks
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant who has been administered a pharmaceutical product. The occurrence, which may or may not have a causal relationship with the investigational treatment, may include any clinical or laboratory change that does not commonly occur in that patient and is considered clinically significant.
Arm/Group | Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg | Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg
All-Cause Mortality (participants affected / at risk) | 6/8 | 3/6
Serious Adverse Events (participants affected / at risk) | 4/8 | 2/6
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg (N=8) | Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg (N=6)
Pneumonia (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 2, Cohort 3: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg (N=8) | Group 2, Cohort 4: Nemvaleukin Alfa 3 mcg/kg + Pembrolizumab 200 mg (N=6)
Pyrexia (General disorders) | 6 | 3
Chills (General disorders) | 4 | 4
Fatigue (General disorders) | 4 | 4
Asthenia (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Swelling (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 3 | 1
Platelet count decreased (Investigations) | 3 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 1
Weight decreased (Investigations) | 2 | 1
White blood cell count decreased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Hypotension (Vascular disorders) | 4 | 1
Hypertension (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 3 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Device occlusion (Product Issues) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT04144517/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT04144517/SAP_001.pdf